CLINICAL TRIAL: NCT06897969
Title: Comparison of Intralesional Triamcinolone and Intralesional Verapamil in the Treatment of Keloids
Brief Title: Comparison of Intralesional Triamcinolone Versus Verapamil for Keloid Treatment
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Dr. Asma Batool, Principal Investigator, Nishtar Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21467/NMU
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Keloid Scars
Keywords: Keloid; Vancouver scar scale; Triamcinolone; Verapamil; Intralesional injection
MeSH Terms: conditions — Keloid | interventions — Triamcinolone Acetonide; Suspensions; Verapamil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verapamil Treatment (Active Comparator): One ml (2.5 mg) of Intralesional Verapamil Injection will be administered monthly. The injections will be administered with an insulin syringe of 27-gauge needle. Administration of the treatment medication will be continued till the keloid is flattened or TOTAL DURATION of three months.
  Interventions: Drug: Verapamil Injection
- Triamcinolone Treatment (Experimental): Intralesional Triamcinolone acetonide (40mg) will be administered monthly. The injections will be administered with an insulin syringe of 27-gauge needle. Administration of the treatment medication will be continued till the keloid is flattened or TOTAL DURATION of three months.
  Interventions: Drug: Triamcinolone Acetonide 1 ml of 40 mg/mL suspension

INTERVENTIONS:
Drug: Triamcinolone Acetonide 1 ml of 40 mg/mL suspension — Monthly intralesional injection
  Arms: Triamcinolone Treatment
Drug: Verapamil Injection — 2.5 mg of intralesional Verapamil injection monthly
  Arms: Verapamil Treatment

SUMMARY:
This study aims to compare the efficacy of intralesional triamcinolone and verapamil in patients presenting with keloid at our local setting. The results will guide us towards better management of keloids by choosing the more appropriate treatment. Adequate treatment will reduce significant emotional and physical distress in patients. We hypothesized that mean reduction in Vancouver Scar Score is higher in triamcinolone acetonide group compared to verapamil after three months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* size of keloid1-5 cm,
* on any site of the body,
* duration less then five years and
* baseline Vancouver scar score of more the or equal to 5

Exclusion Criteria:

* Pregnant or lactating women,
* family history of keloids,
* acromegaly, and
* congestive cardiac diseases

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Vancouver Scar Score | Vancouver Scar score will be measured at baseline (before treatment assignment) and then 4-weeks after completion of treatment - 16-weeks after randomization.
  The Vancouver Scar scale assesses four parameters of vascularity, pigmentation, pliability and height. The total score ranges from 0 - 13.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Aliya Akhtar, FCPS, Study Director — Nishtar Medical University
Locations (1):
- Nishtar Medical University & Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to protect patient confidentiality and comply with ethical and regulatory guidelines. Additionally, the study design does not include provisions for public data sharing.

REFERENCES:
- [Background] Kuang J, An P, Li W. Comparative efficacy and safety of verapamil and triamcinolone in keloid and hypertrophic scar treatment: a meta-analysis. J Cosmet Laser Ther. 2021 Feb 17;23(1-2):26-34. doi: 10.1080/14764172.2021.1950765. Epub 2021 Jul 18. PMID 34278918
- [Background] Uzair M, Butt G, Khurshid K, Pal SS. Comparison of intralesional triamcinolone and intralesional verapamil in the treatment of keloids. Our Dermatol Online. 2015;6(3):280-4.
- [Background] Saki N, Mokhtari R, Nozari F. Comparing the Efficacy of Intralesional Triamcinolone Acetonide With Verapamil in Treatment of Keloids: A Randomized Controlled Trial. Dermatol Pract Concept. 2019 Jan 31;9(1):4-9. doi: 10.5826/dpc.0901a02. eCollection 2019 Jan. PMID 30775139